CLINICAL TRIAL: NCT01067352
Title: An Open, Multicenter, Randomized, Controlled Trial to Evaluate the Correlation Between Spontaneous Catch-up Growth, Clinical Response to Saizen (Recombinant Human Growth Hormone, r-hGH) and Gene Expression Profiling in Children Small for Gestational Age (SGA)
Brief Title: A Trial to Evaluate the Correlation Between Spontaneous Catch-up Growth, Clinical Response to Saizen (Recombinant Human Growth Hormone, r-hGH) and Gene Expression Profiling in Children Small for Gestational Age (SGA)
Acronym: SAIZEN in SGA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was discontinued prematurely due to difficulty in participant recruitment.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.P.A., Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP23681
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Infant, Small for Gestational Age
Keywords: Infant, small for gestational age; Growth hormone; Saizen
MeSH Terms: interventions — Growth Hormone; Human Growth Hormone

ARMS (3):
- Group A (A1) (Experimental): Participants were allocated to Group A if were still third percentile for height (according to the Tanner reference table) at the age of 4-6 years. Group A would be then randomized to receive Saizen at the daily dose of 0.035 milligram (mg)/kilogram (kg) (Group A1) or no treatment (Group A2) for two years.
  Interventions: Drug: Recombinant human growth hormone (r-hGH)
- Group A (A2) (No Intervention): Participants were allocated to Group A if were still third percentile for height (according to the Tanner reference table) at the age of 4-6 years. Group A would be then randomized to receive no treatment (Group A2) for two years.
- Group B (No Intervention): Participants were allocated to Group B being third percentile (thus showing a spontaneous catch-up growth).

INTERVENTIONS:
Drug: Recombinant human growth hormone (r-hGH) — Recombinant human GH were administered subcutaneously (s.c) at the daily dose of 0.067 mg/kg of body weight to Group A1.
  Other Names: Saizen
  Arms: Group A (A1)

SUMMARY:
This open, multicentric, randomized, controlled study is planned to evaluate the correlation between gene expression, spontaneous catch-up growth and therapeutic response to Saizen in SGA children.

DETAILED DESCRIPTION:
This open, multicentric, randomized, controlled study was planned to identify genes activated by hGH in SGA children responders to treatment (making it possible in the near future to better identify SGA children likely to benefit from hGH treatment). Furthermore, the study would hopefully allow to verify which genes were responsible of spontaneous catch-up growth in children with diagnosis of SGA at birth but above the third percentile for height at the age of 24 months, and if these genes were the same activated by hGH during the treatment in participants responders. Sixty children born at term (i.e. after the 37th completed week of gestation) and with a diagnosis of SGA (defined as a length less than tenth percentile according to the Italian reference table published by Bertini and Fabris) were planned to be enrolled in the study. Forty participants (group A) were still less than third percentile for height (according to the Tanner reference table) at the age of 24 months, the remaining 20 (group B) being more than or equal to third percentile (thus showing a spontaneous catch-up growth). Group A was randomized to receive Saizen at the daily dose of 0.067 mg/kg (Group A1) or no treatment (Group A2) for two years. All participants were to undergo full clinical examination and blood chemistry at baseline visit and visit after 1,6,12,18 and 24 months for a period of two years. Gene expression analysis using the Clontech Atlas Human Array was performed in all participants at baseline and after one year in order to identify the possible correlation between catch-up growth (either spontaneous or drug-induced) and expression of some genes.

OBJECTIVES

Primary objective:

* To evaluate the correlation between gene expression profiling and catch-up growth (either spontaneous or drug induced after one year of treatment) in SGA children.

Secondary Objectives:

* To evaluate the percentage of participants not treated who show a spontaneous catch-up growth during the two years of observation.
* To assess the safety and tolerability of early treatment with Saizen

ELIGIBILITY:
Inclusion Criteria:

* SGA at birth (defined as a length at birth equal or below the tenth percentile according to the Italian reference table of Bertini and Fabris)
* Age of 24 Months
* Caucasic
* Born at term (i.e. after the 37th completed week of gestation)
* Height equal or below (Group A) or up (Group B) the third percentile at the age of 24 months according to the Tanner reference table
* Sufficient GH secretion (more than 10 nanogram (ng)/milliliter (ml)) at least to one of the tests commonly used at that age (glucagon, Levo-dopa, arginine, clonidine, Growth Hormone Releasing Hormone (GHRH), GH integrated secretion)
* Normal level of Thyroid-stimulating hormone (THS), Free Triiodothyronine (FT3), Free Thyroxine (FT4), Insulin-like growth factor 1(IGF-1), insulin and haemoglobin A1c (HbA1c)
* Normal level of Immunoglobulin A (IgA)
* Children parents willing to comply with the protocol for the whole duration of the study
* A written Informed Consent before the baseline visit must be obtained from the parent(s) / legal guardian(s)

Exclusion Criteria:

* Congenital malformations (including Silver-Russel syndrome)
* Known abnormal karyotype, especially in girls
* Twins
* Severe psychomotor retardation
* Previous or ongoing treatment with anabolic steroids or r-hGH
* Treatments interfering with the immune system (including bacterial lysate)
* Severe chronic illnesses
* Autoimmune diseases

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2004-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.P.A., Italy
Locations (1):
- Merck Serono S.p.A., Roma, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 12 study centers in Italy from 20 Feb 2004 to 10 Jul 2009.
Groups:
- Group A, Less Than Third Percentile (Saizen): Participants with less than third percentile for height (according to the Tanner reference table) at the age of 4-6 years received Saizen (recombinant human growth hormone, r-hGH) subcutaneously (s.c) at the daily dose of 0.035 milligram(mg)/kilogram(kg) for 2 years.
- Group A2, Less Than Third Percentile (No Treatment): Participants with less than third percentile for height (according to the Tanner reference table) at the age of 4-6 years received no drug treatment for 2 years.
- Group B, More Than Third Percentile (No Treatment): Participants with more than third percentile for height (according to the Tanner reference table) at the age of 4-6 years received no drug treatment for 2 years.
Period: Overall Study
Arm/Group | Group A, Less Than Third Percentile (Saizen) | Group A2, Less Than Third Percentile (No Treatment) | Group B, More Than Third Percentile (No Treatment)
Started | 9 | 6 | 10
Completed | 8 | 3 | 9
Not Completed | 1 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A, Less Than Third Percentile (Saizen) | Group A2, Less Than Third Percentile (No Treatment) | Group B, More Than Third Percentile (No Treatment) | Total
Number analyzed (Participants) | 9 | 6 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.7 (1.2) | 5.0 (0.7) | 5.2 (0.4) | 5.3 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 5 | 2 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Gene Expression Profiling and Catch-up Growth in Small for Gestational Age (SGA) Children
Description: Gene expression profiling:analysis of ribonucleic acid (RNA) extracted from body tissue or fluids using Clontech Atlas Human Array to study level of activation of genes in tissue analyzed. Analysis was performed to identify possible correlation between catch-up growth (either spontaneous or drug-induced after Week 48) and therapeutic response to rhGH. Spontaneous catch up growth:shown by SGA participants having length more than third percentile at Week 96 without any treatment;drug induced growth was by SGA participants having length more than third percentile at Week 96 with drug treatment.
Time Frame: Baseline and Week 48
Population: Gene expression profiling was not performed due to RNA degradation in nearly all of the blood samples and hence no comparison between gene expression and growth was made.
Arm/Group | Group A, Less Than Third Percentile (Saizen) | Group A2, Less Than Third Percentile (No Treatment) | Group B, More Than Third Percentile (No Treatment)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Untreated Participants Who Showed a Spontaneous Catch-up Growth
Description: Spontaneous catch up growth was the growth shown by SGA participants having length more than third percentile at Week 96 without any study drug treatment.
Time Frame: Baseline through Week 96
Population: Data was not analyzed due to small number of evaluable participants.
Arm/Group | Group A, Less Than Third Percentile (Saizen) | Group A2, Less Than Third Percentile (No Treatment) | Group B, More Than Third Percentile (No Treatment)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Study Drug Discontinuation
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug , SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued from the study due to AE were also recorded.
Time Frame: Baseline through Week 96
Population: Safety analysis population included all randomized participants with at least 1 post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | Group A, Less Than Third Percentile (Saizen) | Group A2, Less Than Third Percentile (No Treatment) | Group B, More Than Third Percentile (No Treatment)
Number analyzed (Participants) | 8 | 4 | 10
participants
  AEs | 6 | 4 | 9
  SAEs | 0 | 0 | 0
  Discontinuation due to AEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected on an ongoing basis from day of written informed consent. All new AEs were recorded until the post-treatment safety, on Day 30 post-drug administration.
Arm/Group | Group A, Less Than Third Percentile (Saizen) | Group A2, Less Than Third Percentile (No Treatment) | Group B, More Than Third Percentile (No Treatment)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 6/8 | 4/4 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A, Less Than Third Percentile (Saizen) (N=8) | Group A2, Less Than Third Percentile (No Treatment) (N=4) | Group B, More Than Third Percentile (No Treatment) (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (15) | 2 (6) | 4 (6)
Ear infection (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (4) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipoprotein (a) abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood insulin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary and secondary efficacy objectives were not met because of poor participant enrollment and no quality RNA samples obtained to evaluate (RNA degradation in nearly all of the blood samples).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other